CLINICAL TRIAL: NCT07174128
Title: Effect of Two Cut-Off Values of Plethysmographic Variability Index to Guide Intraoperative Fluid Therapy on Serum Lactate in Patients Undergoing Excision of Supra-Tentorial Brain Tumors: A Randomized Controlled Study
Brief Title: Two Cut-Off Values of Plethysmographic Variability Index to Guide Intraoperative Fluid Therapy on Serum Lactate in Patients Undergoing Excision of Supra-Tentorial Brain Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelrahman Gomaa Abdelhameed Eltokhy, Assistant Lecturer of Anesthesia, Pain Management and surgical ICU, Faculty of Medicine, Cairo University, Cairo, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD--452-2023
Record Dates: First submitted 2025-09-04; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cut-Off Value; Plethysmographic Variability Index; Intraoperative; Fluid Therapy; Serum Lactate; Excision; Supra-Tentorial Brain Tumors
MeSH Terms: interventions — Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low PVI group (Experimental): Patients would receive the second round of fluid loading if the Plethysmographic Variability Index (PVI) was 14%.
  Interventions: Other: Fluid Therapy
- High PVI gro (Experimental): Patients would receive the second round of fluid loading if the Plethysmographic Variability Index (PVI) was 20%.
  Interventions: Other: Fluid Therapy

INTERVENTIONS:
Other: Fluid Therapy — Patients would receive the second round of fluid loading if the Plethysmographic Variability Index (PVI) was 14%.
  Arms: Low PVI group
Other: Fluid Therapy — Patients would receive the second round of fluid loading if the Plethysmographic Variability Index (PVI) was 20%.
  Arms: High PVI gro

SUMMARY:
This study aimed to compare two cut-off values of plethysmographic variability index (PVI) -guided fluid therapy in patients undergoing supra-tentorial mass excision regarding immediate postoperative serum lactate.

DETAILED DESCRIPTION:
Fluid therapy in patients undergoing craniotomy is very critical; hypovolemia might decrease cerebral perfusion, while fluid overinfusion might cause brain swelling that impairs surgical removal of lesions.

The plethysmographic variability index (PVI) is one of the dynamic indices of fluid responsiveness, a simple, automatic, non-invasive, and continuous method based on calculating changes in the perfusion index (PI).

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old.
* Both sexes.
* Patients scheduled for supra-tentorial brain tumor excision.

Exclusion Criteria:

* Arrhythmias.
* Pulmonary hypertension.
* Impaired cardiac contractility.
* Impaired liver or kidney function.
* Low lung compliance.
* Body mass index above 40.
* Intra-operative hemodynamic instability on vasopressors or inotropes.
* Peripheral arterial occlusive diseases.
* Hand injuries or burns that preclude the application of the Masimo device probe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-08-24 (Actual); Study Completion 2025-08-24 (Actual)

PRIMARY OUTCOMES:
Serum lactate level | 24 hours postoperatively
  Serum lactate level was measured at the end of surgery (immediately after extubation).

SECONDARY OUTCOMES:
Brain Relaxation scale | Intraoperatively
  The neurosurgeon assessed the Brain Relaxation scale at three time intervals: with dural opening, after two hours, and before dural closure. A 4-point scale will be performed as follows: grade 1, perfectly relaxed; grade 2, satisfactorily relaxed; grade 3, firm brain; grade 4, bulging brain.
Heart rate | 20 minutes after fluid loading
  Heart rate was measured immediately after fluid loading and every 5 minutes for 20 minutes.
Mean arterial pressure | 20 minutes after fluid loading
  Mean arterial pressure was measured immediately after fluid loading and every 5 minutes for 20 minutes.
Length of hospital stay | Till discharge from the hospital (Up to 2 weeks)
  Length of hospital stay was recorded from admission till discharge from the hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.